CLINICAL TRIAL: NCT05180942
Title: Statins and prOgression of Coronary atheRosclerosis in melanomA Patients Treated With chEckpoint inhibitorS
Acronym: SOCRATES
Status: Recruiting | Type: Observational
Sponsor: Monash University (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Stephen Nicholls, Professor, Monash University
Other Study IDs: SOCRATES
Record Dates: First submitted 2021-11-11; First posted 2022-01-06 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Melanoma; Atherosclerosis
MeSH Terms: conditions — Melanoma; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional blood samples will be collected for Future Biomedical Research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is a prospective observational study evaluating the natural history of coronary plaque burden in participants with melanoma treated with ICI. The study will be conducted at various sites across Australia.

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing informed consent and willing to adhere to all protocol requirements
* patients aged > or equal to 40 years
* Histologically confirmed melanoma of any stage planned for, commenced, or completed treatment with ICI
* having acceptable imaging quality deemed by the core laboratory
* Investigator believes that the participant is willing to adhere to all protocol requirements, including returning for follow up CTCA.

Exclusion Criteria:

* Known clinically manifest cardiovascular disease
* Female participants must not be pregnant, breastfeeding or plan to become pregnant during the study.
* Estimated glomerular filtration rate of <45 mL/min calculated using the Chronic Kidney Disease Epidemiology Collaboration equation
* Severe liver disease or cirrhosis
* History of any other malignancy within the past 5 years in addition to melanoma with the exception of non-melanoma skin cancers
* Prognostic factors associated with an expected survival less than 18 months at Investigators' discretion (e.g. unresectable brain metastases)
* Evidence of any other clinically significant non-cardiac disease or condition that, in the opinion of the Investigator, would preclude participation in the study
* Major allergy to iodine
* Participation in another clinical trial that does not allow participation in multiple trials at the same time

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 40 years and older with melanoma of any stage, who are planned for, currently receiving or have received treatment with an ICI may be considered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To determine the natural history of the burden and composition of coronary atherosclerosis in individuals with melanoma treated with ICIs. | 18 months
  The change in non-calcified coronary plaque volume will be measured on serial computed tomography coronary angiography scans.

SECONDARY OUTCOMES:
To determine the prevalence of CV risk factors in individuals with melanoma treated with ICIs. | 18 months
To determine the relationship between statin use and the burden, composition and progression of coronary atherosclerosis in individuals with melanoma treated with ICIs. | 18 months
  The change in non-calcified coronary plaque volume as measured on serial computed tomography coronary angiography scans will be compared between patients treated with statins and patients not treated with statins in the study.
To examine the impact of using CTCA to guide preventative therapy with statins in patients with melanoma treated with ICIs. | 18 months
  The number of patients who were started on statin therapy by their treating clinicians after undergoing computed tomography coronary angiography in the study will be recorded.
To evaluate the impact of participation in a cardio-oncology trial on measures of quality of life in patients with melanoma treated with ICIs. | 18 months
  Quality of life will be assessed by using the PHQ-9, GAD-7, EORTC QLQ-C30, EuroQOL EQ-5D, and FACT-M questionnaires at baseline and at 18 month follow up. The change in quality of life scores on each questionnaire will be compared with historical cohorts that have previously been reported in the literature.
To determine the incidence of major atherosclerotic cardiovascular events in patients with melanoma treated with ICIs. | 18 months
To determine progression free survival with regard to the underlying melanoma following treatment with ICIs. | 18 months
To determine overall survival in patients with melanoma treated with ICIs. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Nicholls, MBBS, PhD, Principal Investigator — Monash University
Locations (12):
- Australia (12):
  - Nepean Hospital, Kingswood, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Bundaberg Base Hospital, Bundaberg, Queensland
  - Hervey Bay Hospital, Hervey Bay, Queensland
  - Ipswich Hospital, Ipswich, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Queen Elizabeth Hospital, Woodville South, South Australia
  - Monash Health, Clayton, Victoria
  - Peninsula Health, Frankston, Victoria
  - Cabrini Health, Malvern, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Mildura Public Base Hospital, Mildura, Victoria

IPD SHARING:
Plan to Share IPD: No
The Steering Committee will decide if and how IPD will be shared. It is expected that study Co Investigators will be able to access data once the primary results have been presented.